CLINICAL TRIAL: NCT03839511
Title: Use of a Hyperinsulinemic-hypyglycemic Clamp to Study Hypoglycemia: a Method Development Study
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, David McDougal, Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: 2018-050-PBRC HYPOCLAMP
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hyperinsulinemic-hypoglycemic clamp — Subjects will arrive at the inpatient unit in the morning after at least a 10 hour overnight fast. Upon arrival to PBRC, participants will be admitted to the inpatient unit. Following measurement of weight, vitals, and pregnancy test (women only), the 4-hour hypoglycemic clamp procedure (30 minute baseline, 120 minute insulin infusion, and 90 minute recovery) will be performed. Upon completion of the clamp procedure, participants will be provided lunch (Standard American Diet). Following lunch, the CGM sensor will be removed and pending a stable blood glucose level in the normal range, the participant will be discharged from the inpatient unit. This completes the study.

SUMMARY:
A hyperinsulinemic-hypoglycemic clamp is an experimental procedure, which allows for hypoglycemia to be studied in a safe and controlled manner. The goal of this study is to establish the hyperinsulinemic-hypoglycemic clamp procedure at Pennington Biomedical Research Center in order to apply the knowledge gained to future studies which will determine the efficacy of our biomarker for predicting susceptibility to hypoglycemia. Additionally, our use of continuous glucose monitoring (CGM) during the clamp procedure will provide novel data regarding the accuracy of CGM during hypoglycemic conditions in a controlled research setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Ages 18-40 years
* BMI between 20 kg/m2 and 30 kg/m2 (±0.5 kg/m2 will be accepted)
* Medically cleared for participation in the study

Exclusion Criteria:

* History of clinically diagnosed diabetes or a fasting blood glucose >126 mg/dL
* Average screening blood pressure >140/90 mmHg
* History of cardiovascular disease
* Pregnant, planning to become pregnant, or breastfeeding
* Based on the investigative team's clinical judgement, a subject may not be appropriate for participation in the study.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: We will enroll up to 8 healthy men or women (goal n=3 completers) in this method development study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants will undergo a hyperinsulinemic-hypoglycemic clamp procedure
Period: Overall Study
Arm/Group | Intervention
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Intervention
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Fasting blood glucose [Mean (Standard Deviation); unit: mg/dL] — Overnight fasting blood glucose at screening
  mg/dL | 86 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Peak Epinephrine Levels
Description: This value represents the average peak epinephrine value measured during the hypoglycemic clamp procedure
Time Frame: 90 minute interval following initiation of insulin infusion
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intervention
Number analyzed (Participants) | 4
pg/mL | 609 (280)

2. Secondary Outcome: CGM Glucose
Description: This value represents the average glucose values measured via continuous glucose monitoring during the hypoglycemic clamp procedure
Time Frame: 90 minute interval following initiation of insulin infusion
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention
Number analyzed (Participants) | 4
mg/dL | 56 (3.9)

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03839511/Prot_000.pdf